CLINICAL TRIAL: NCT01417650
Title: A Randomized Clinical Trial of the Effect of Low Level Laser Therapy on Improvement of Temporomandibular Joint Osteoarthritis
Brief Title: The Effect of Low Level Laser Therapy on Improvement of Temporomandibular Joint Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Azam Madani, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 89342
Record Dates: First submitted 2011-08-08; First posted 2011-08-16 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2010-06

CONDITIONS: Temporomandibular Joint Disorder
Keywords: temporomandibular disorder; laser therapy; osteoarthritis
MeSH Terms: conditions — Temporomandibular Joint Disorders; Osteoarthritis | interventions — Low-Level Light Therapy; Laser Therapy; Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laser (Active Comparator): In this group, the 890 nm diode laser (Mustang 2000+,Russia) will be used with frequency of 1500 Hz, and dose of 2 J/cm2 per point in the joint area and painful muscles if any.
  Interventions: Radiation: Low level laser therapy
- placebo (Placebo Comparator): In this group the low power laser will be applied with minimal dose that is very lower than the threshold necessary for therapeutic effects.
  Interventions: Radiation: Low level laser therapy

INTERVENTIONS:
Radiation: Low level laser therapy — In this group, the 890 nm diode laser (Mustang 2000+, Russia) will be applied with frequency of 1500 Hz, and dose of 2 J/cm2 per point in the joint area and painful muscles if any.
  Other Names: low power laser, laser therapy, diode laser
  Arms: laser
Radiation: Low level laser therapy — In this group, the low level laser will be applied with a minimal dose that is very lower than the threshold necessary for therapeutic effects.
  Other Names: low power laser, laser therapy, diode laser
  Arms: placebo

SUMMARY:
Temporomandibular disorder (TMD) is the major cause of nondental pain in orofacial area. Laser therapy can be considered as one of the most popular methods of pain relief in TMD patients. The special features of laser light such as coherence, monochromaticity, and collimation can result in the ability of laser light to modify cellular metabolism, increase tissue repair and reduce edema and inflammation. The effectiveness of low level laser therapy in reducing the signs and symptoms of temporomandibular joint disorders has been investigated in a few studies. But, in most of the previous studies the etiology of TMD has not been considered in patient selection. Furthermore, there are some controversies in the results of these studies. According to our data, there is no study evaluating the effects of low level laser therapy on patients having TMJ osteoarthritis.

The aim of this study is to evaluate the effectiveness of low level laser therapy in improving osteoarthritis of temporomandibular joint and also to evaluate the long term effects of laser therapy on the morphology of the joint.

DETAILED DESCRIPTION:
Project method: This study will be implemented on 20 patients aged 35-60 years referring to Department of Prosthetic Dentistry of Mashhad Dental School. The patients are selected according to the RDC/TMD criteria to include those having temporomandibular osteoarthritis with unknown etiology. The patients will be asked to take cone beam CT of temporomandibular joint to evaluate any changes in morphology of the TMJ. The patients will be randomly assigned to two groups: Group 1 (treatment group) will receive low level laser therapy. The laser light will be applied with 890 nm diode laser (Mustang 2000+, Russia) with frequency of 1500 Hz, and dose of 2 J/cm2 per point in the joint area and painful muscles if any. In Group 2 (placebo) the low power laser will be applied with a minimal dose that is very lower than the threshold necessary for therapeutic effects. Laser therapy for both the treatment and placebo groups will be applied in the back, front, and above the mandibular condyles and inside the external auditory meatus and also on painful muscles three times a week for four weeks. Patients will be evaluated at the start of the treatment, after the 6th and 12th sessions of laser therapy and also one month after the end of the treatment. At each evaluation, the pain level in opening the mouth and masticatory muscle tenderness will be measured according to the Visual Analogue Scale (VAS). The range of lateral and protrusive mandibular movements, the difficulty in chewing food and the the presence or absence of sound joints will also be evaluated. One year after treatment, the patients will be referred for taking the second cone beam CT of the TMJ to seek any change in morphology of the joint.

ELIGIBILITY:
Inclusion Criteria:

* The patients are selected according to the RDC/TMD criteria to include those having temporomandibular osteoarthritis with unknown etiology.

Exclusion Criteria:

1. Patients with systemic problems.
2. Patients using analgesic or antidepressant drugs.
3. Patients undergoing any treatment modality for TMD disease.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-10 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Pain relief | Up to 1 month after laser theray
  Pain is assessed by visual analogue scale (VAS)

SECONDARY OUTCOMES:
TMD sounds | Up to 1 month after laser therapy
  The presence or absence of articular sounds is checked.
Mouth opening measurement | Up to 1 month after laser therapy
  The amount of mouth opening with and without pain is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Farzaneh Ahrari, DDS, MS, Principal Investigator — Mashhad University of Medical Sciences